CLINICAL TRIAL: NCT03718559
Title: A Multi-centre, Open-labelled, Randomized Controlled Trial Comparing Two Different Anticoagulation Strategies in High-risk Atrial Fibrillation and Stable Coronary Artery Disease
Brief Title: Edoxaban Versus Edoxaban With antiPlatelet Agent In Patients With Atrial Fibrillation and Chronic Stable Coronary Artery Disease
Acronym: EPIC-CAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gi-Byoung Nam (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Gi-Byoung Nam, Professor, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCVEP2018-01
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease; Stable Angina; Stable Chronic Angina
Keywords: Edoxaban; antiplatelet; anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease; Angina, Stable | interventions — edoxaban; Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban alone (Experimental)
  Interventions: Drug: Edoxaban Monotherapy
- Combination of edoxaban plus single antiplatelet (Active Comparator)
  Interventions: Drug: Edoxaban plus Single Antiplatelet Agent

INTERVENTIONS:
Drug: Edoxaban Monotherapy — Taking edoxaban (Lixiana™, Daiichi-Sankyo Inc.) 60mg once daily. The dose of edoxaban will be reduced to 30mg once daily in patients with estimated creatinine clearance 15≤CrCL≤50mL/min by Cockcroft-Gault equation or weight is ≤60kg.
  Other Names: Lixiana™
  Arms: Edoxaban alone
Drug: Edoxaban plus Single Antiplatelet Agent — Type of antiplatelet agent is dependant upon the investigator's discretion, but aspirin 100mg once daily or clopidogrel 75mg once daily was recommended.
  Arms: Combination of edoxaban plus single antiplatelet

SUMMARY:
This study evaluates the efficacy and safety of Edoxaban with the combination of edoxaban and antiplatelet in patients with stable CAD (coronary artery stenosis ≥50% on medical treatment or revascularized stable CAD [≥ 12 months for acute coronary syndrome and ≥ 6 months after stable CAD]) and high-risk atrial fibrillation (CHA2DS2-VASc score ≥2).

ELIGIBILITY:
Inclusion Criteria

1. A subject was ≥ 18 years of age
2. Patients with nonvalvular atrial fibrillation with high embolic risk (CHA2DS2-VASc score ≥2)
3. Patients with Stable coronary artery disease

   * Anatomically confirmed coronary artery disease (with ≥50% stenosis of major epicardial coronary artery documented by cardiac catheterization or coronary computed tomographic angiography) on medical therapy alone.
   * Revascularized coronary artery disease (either Percutaneous Coronary Intervention or coronary bypass surgery) whom the last revascularization should be performed ≥12 months before study enrollment for the acute coronary syndrome and ≥6 months for stable angina pectoris.

Exclusion Criteria

1. Patients with thrombocytopenia
2. High risk of bleeding which prohibits the anticoagulant use. (baseline comorbidities, hyper or hypercoagulable state, increased prothrombin time or activated partial thromboplastin time)
3. Prior history of intracranial haemorrhage
4. Mechanical prosthetic valve or moderate to severe mitral stenosis
5. The risk of bleeding increased due to the following reasons;

   * i. history of gastrointestinal ulcers within 1 month
   * ii. Malignant tumor with high risk of bleeding
   * iii. Brain or spinal cord injury within 1 month
   * iv. History of intracranial or intracerebral hemorrhage within 12 months
   * v. Esophageal varices
   * vi. Spinal cord vascular abnormalities or intracerebral vascular abnormalities
   * vii. Active bleeding
   * viii. Hemoglobin level <7.0 g/dL or platelet count ≤ 50,000 / mm3
   * ix. History of major surgery within 1 month
6. Uncontrolled severe hypertension
7. Hemodynamically Unstable or pulmonary embolism requiring thrombolysis or pulmonary embolectomy
8. History of hypersensitivity to Edoxaban, aspirin, or clopidogrel
9. Genetic problem with galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
10. Planned Percutaneous Coronary Intervention or coronary bypass surgery was planned within 1 year after randomization
11. Liver cirrhosis or liver dysfunction (AST or ALT > x3 of normal range or coagulation abnormality)
12. Estimated CrCl by Cockcroft-Gault equation<15 mL/min
13. Life expectancy less than 12 months
14. The subject was unable to provide written informed consent or participate in long-term follow-up
15. Pregnant and/or lactating women
16. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Rate of net Clinical Outcome | 1 year
  composites of death, stroke, systemic embolic event, myocardial infarction, unplanned revascularization of a major coronary artery, major bleeding, and clinically relevant non-major bleeding event

SECONDARY OUTCOMES:
Rate of all cause death | 1 year
Rate of cardiovascular death | 1 year
Rate of myocardial infarction | 1 year
Rate of ischemic stroke | 1 year
Rate of systemic embolism | 1 year
Rate of unplanned revascularization | 1 year
Rate of composite of hard outcomes | 1 year
  all cause death, myocardial infarction, ischemic stroke, and systemic embolism
Rate of stent thrombosis | 1 year
Rate of composite of Major or clinically relevant non-major bleeding | 1 year
  1. Major bleeding
     * Fatal bleeding
     * Bleeding in the critical site (Intracranial, retroperitoneal, intraocular, intraspinal, intra-articular, pericardial, intramuscular with compartment syndrome)
     * Bleeding causing a fall in haemoglobin level of 2g/dL or leading to transfusion of two or more units of whole blood or red cells.
  2. Clinically relevant non-major bleeding
  defined as any sign or symptom of haemorrhage that does not fit the criteria for The International Society on Thrombosis and Haemostasis (ISTH) major bleeding but requiring medical intervention, leading to hospitalization, or prompting a medical evaluation. Specifically bleeding that meet one of following criteria.
  * bleeding that resulted in hospitalization
  * medical or surgical intervention for bleeding
  * an unscheduled clinic visit, or
  * a change in physician-directed antithrombotic therapy.
Rate of fatal bleeding | 1 year
  International Society on Thrombosis and Haemostasis(ISTH), The Bleeding Academic Research Consortium (BARC)5
Rate of major bleeding | 1 year
  ISTH, BARC 3, The Thrombolysis in Myocardial Infarction (TIMI) major bleeding
Rate of minor bleeding | 1 year
  ISTH, BARC and TIMI criteria
Rate of intracranial hemorrhage | 1 year
Rate of gastrointestinal hemorrhage | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Duk-woo Park, MD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (18):
- South Korea (18):
  - Hallym University Medical Center, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Dongguk University Ilsan Hospital, Ilsan
  - Dong-A University Hospital, Pusan
  - Inje University Haeundae Paik Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Kangdong KyungHee University hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic Univ. of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic Univ.of Korea Eunpyeong St.Mary's Hospital, Seoul
  - VHS medical center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Ulsan Univeristy Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho MS, Kang DY, Lee JB, Oh YS, Lee CH, Choi EK, Lee JH, Kwon CH, Park GM, Choi HO, Park KH, Park KM, Hwang J, Yoo KD, Cho YR, Kim JH, Hwang KW, Jin ES, Kwon O, Kim KH, Park DW, Nam GB; on the behalf of the EPIC-CAD Investigators. Off-label underdosing of edoxaban antithrombotic therapy for patients with atrial fibrillation and stable coronary artery disease: findings from the EPIC-CAD trial. Heart. 2025 Sep 9:heartjnl-2025-326646. doi: 10.1136/heartjnl-2025-326646. Online ahead of print. PMID 40930594
- [Derived] Cho MS, Kang DY, Ahn JM, Yun SC, Oh YS, Lee CH, Choi EK, Lee JH, Kwon CH, Park GM, Choi HO, Park KH, Park KM, Hwang J, Yoo KD, Cho YR, Kim JH, Hwang KW, Jin ES, Kwon O, Kim KH, Park SJ, Park DW, Nam GB; EPIC-CAD Investigators. Edoxaban Antithrombotic Therapy for Atrial Fibrillation and Stable Coronary Artery Disease. N Engl J Med. 2024 Dec 5;391(22):2075-2086. doi: 10.1056/NEJMoa2407362. Epub 2024 Sep 1. PMID 39225258